CLINICAL TRIAL: NCT04160130
Title: A Prospective, Randomized, Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Transcatheter Aortic Valve Implantation in Female Patients Who Have Severe Symptomatic Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: RHEIA (Randomized researcH in womEn All Comers With Aortic Stenosis)
Acronym: RHEIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Optimapharm (Industry)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RHEIA; CIV-19-11-030544 (Other: DIMDI)
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
Keywords: Research in woman; Transcatheter Aortic Valve Implantation (TAVI); surgical aortic valve replacement (SAVR); cardiovascular disease; heart disease; Sapien 3; Transcatheter Aortic Valve Replacement (TAVR)
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Cardiovascular Diseases; Heart Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAPIEN 3 or SAPIEN 3 Ultra (Experimental): Edwards SAPIEN 3 THV system Model 9600 TFX (20, 23, 26 and 29 mm) or SAPIEN 3 Ultra THV system Model 9750 TFX (20, 23, 26) with the associated transfemoral delivery systems.
  Interventions: Procedure: Transcatheter aortic valve replacement
- any surgical bioprosthetic aortic valve (Active Comparator): Any commercially available surgical bioprosthetic valve
  Interventions: Procedure: Transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — Patients will be randomized 1:1 to receive either transcatheter aortic valve replacement (TAVI) or aortic valve replacement with a commercially available surgical bioprosthetic valve.
  Other Names: Surgical aortic valve replacement

SUMMARY:
Purpose of this prospective, randomized, controlled, multi-center study is to evaluate the safety and efficacy of Transcatheter Aortic Valve Implantation (TAVI) as compared to surgical aortic valve replacement (SAVR) in female patients with severe symptomatic aortic stenosis. Patients will be randomized 1:1 to receive either TAVI or SAVR aortic valve replacement. For TAVI procedure, Edwards SAPIEN 3 THV system Model 9600 TFX (20, 23, 26 and 29 mm) or SAPIEN 3 Ultra THV system Model 9750 TFX (20, 23, 26) with the associated transfemoral delivery systems will be sued, for SAVR any commercially available surgical bioprosthetic valve. Patients will undergo the following visits: Screening, Procedure, Post Procedure, Discharge, 30 day, 6 months (telephone contact) and 1 year.

DETAILED DESCRIPTION:
Recent large meta-analyses and a large retrospective study from the STS/ACC TVT Registry demonstrated improved survival in female versus male aortic sclerosis patients undergoing TAVI despite their advanced age and increased rates of major peri-procedural vascular complications, bleeding events and strokes. These gender-related patient profile differences have also been present in multicentre cohorts across the world. A recent meta-analysis by Siontis et al. showed that TAVI, when compared with SAVR, was associated with a significant 13% relative risk reduction in 2-year mortality, a benefit more pronounced amongst females and patients undergoing transfemoral TAVI.

In a recent meta-analysis, the female-specific survival advantage from TAVI over SAVR was explored. Amongst females, TAVI recipients had a significantly lower mortality than SAVR recipients, at 1 year (OR 0.68; 95%CI 0.50 to 0.94). Amongst males there was no difference in mortality between TAVI and SAVR at 1 year (OR 1.09; 95%CI 0.86 to 1.39). There was statistically significant evidence of a difference in treatment effect between genders at 1 year (p interaction = 0.02). In an attempt to explore the mechanisms for an increased mortality rate in women undergoing SAVR, different endpoints were explored in female patients exclusively. It was shown that women, undergoing SAVR, having both a higher periprocedural mortality, higher rates of bleeding and acute kidney injury, worse patient prosthesis match and worse long term recovery of left ventricular function.In the recent PARTNER 3 the composite of death from any cause, stroke, or rehospitalization had occurred in 42 patients (8.5%) in the TAVI group as compared with 68 patients (15.1%) in the surgery group at 1 year. The difference was 6.6% (95%CI -10.8% to -2.3%) and thus exceeded the pre-defined non-inferiority margin of 6%.

Subgroup analyses of the primary end point at 1 year showed no heterogeneity of treatment effect in any of the subgroups that were examined including gender (p=0.27). There were 292 women included with an endpoint rate of 18.5% for SAVR (men 13.8%) and 8.1% for TAVI (men 8.7%), showing a clear trend for an increased benefit of women undergoing TAVI instead of SAVR (rate difference -10.4%; 95%CI -18.3% to -2.5%). Nonetheless, the benefits of TAVI were preserved in both men and women.Earlier observational and clinical studies indicated an increased risk for women undergoing SAVR compared to men while being at a comparable risk for TAVI. In a recent meta-analysis of TAVI vs. SAVR in men and women the risk of dying from the intervention was reduced by a relative 32% in women (OR 0.38; 95%CI 0.50-0.94) while there was no such difference in men (OR 1.09; 95%CI 0.86-1.39). This was mostly documented as being the effect of a reduced periprocedural mortality with TAVI (-54%; OR 0.46; 95%CI 0.22-0.96) and major bleeding (-57%; OR 0.43; 95%CI 0.25-0.73) while the difference in strokes and acute kidney injury did not reach statistical significance. Taken all available scientific data on the comparison of TAVI versus open surgery in patients with indication for AVR together it remains probable, that independently of the individual surgical risk female patients in particular seem to benefit from a non-surgical aortic valve replacement strategy.

As the indirect comparisons of the intermediate to low risk outcomes in PARTNER 2/3 suggest a favorable risk reduction in women compared to men as described, the investigators believe it is timely for a dedicated trial to demonstrate the non-inferiority of TAVI in women compared to SAVR and, in case of this being true, whether TAVI is actually superior to performing SAVR.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with severe aortic stenosis as follows:

   • High gradient severe AS (Class I Indication for aortic valve replacement [AVR]): Jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg with Aortic Valve Area (AVA) ≤ 1.0 cm^2 or AVA index ≤ 0.6 cm^2/m^2 OR

   • Low gradient severe aortic stenosis (Class I/IIa indication of AVR) Jet velocity < 4.0 m/s and mean gradient < 40 mmHg and AVA ≤ 1.0 cm^2 and AVA index ≤ 0.6 cm^2/m^2 with confirmation of severe AS by: mean gradient ≥40 mmHg on dobutamine stress echocardiography and/or aortic valve calcium score ≥ 1200 AU on non-contrast CT.

   AND
   * NYHA Functional Class ≥ II OR
   * Exercise test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia
2. Age ≥ 18 years
3. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

1. Patient is not a candidate for both surgical and transcatheter aortic valve replacement.
2. Native aortic annulus size unsuitable for sizes 20, 23, 26, or 29 mm THV based on 3D imaging analysis
3. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
4. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before randomization
5. Aortic valve is unicuspid, bicuspid, or is non-calcified
6. Severe aortic regurgitation (>3+)
7. Any concomitant valve disease that requires an intervention
8. Pre-existing mechanical or bioprosthetic valve in any position (mitral ring is not an exclusion).
9. Complex coronary artery disease:

   * Unprotected left main coronary artery stenosis
   * Syntax score > 32 (in the absence of prior revascularization)
   * Heart Team assessment that optimal revascularization cannot be performed.
10. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days before randomization
11. Leukopenia (WBC < 3000 cell/mcL), anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mcL), history of bleeding diathesis or coagulopathy, or hypercoagulable states
12. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days before randomization
13. Hypertrophic cardiomyopathy with obstruction
14. Ventricular dysfunction with lleft ventricular ejection fraction < 30%
15. Cardiac imaging (echo, CT, and/or MRI) evidence of intracardiac mass, thrombus or vegetation
16. Inability to tolerate or condition precluding treatment with anti- thrombotic/anticoagulation therapy during or after the valve implant procedure
17. Stroke or transient ischemic attack within 90 days before randomization
18. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy
19. Active bacterial endocarditis within 180 days of randomization
20. Severe lung disease (FEV1 < 50%) or currently on home oxygen
21. Severe pulmonary hypertension (e.g., pulmonary arterial systolic pressure ≥ 2/3 systemic pressure)
22. History of cirrhosis or any active liver disease
23. Significant abdominal or thoracic aortic disease (such as porcelain aorta, aneurysm, severe calcification, aortic coarctation, etc.) that would preclude safe passage of the delivery system or cannulation and aortotomy for surgical AVR.
24. Hostile chest or conditions or complications from prior surgery that preclude safe reoperation (e.g., mediastinitis, radiation damage, abnormal chest wall, adhesion of aorta or internal mammary artery to sternum, etc.)
25. Patient refuses blood products
26. BMI > 50 kg/m^2
27. Estimated life expectancy < 24 months
28. Absolute contraindications or allergy to iodinated contrast agent that cannot be adequately treated with pre-medication
29. Immobility that would prevent completion of study procedures
30. Currently participating in an investigational drug or another device study.
31. Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 432 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  Number of patients with death of any cause (death due to proximate cardiac cause, death caused by non-coronary vascular conditions, procedure-related deaths, valve-related deaths, sudden or unwitnessed death, non-cardiovascular mortality, death of unknown cause)
Stroke | through study completion, an average of 1 year
  Number of patients with stroke (disabling and non-disabling).
Re-hospitalization | through study completion, an average of 1 year
  Number of patients with re-hospitalization (valve-related or procedure-related or worsening of congestive heart failure).

SECONDARY OUTCOMES:
Length of Index hospitalization | through day of procedure until day of discharge
  Number of days per patient for index hospitalization.
Prosthesis-patient mismatch | up to 30 days post-procedure
  Number of patients with a prosthesis mismatch.
New onset atrial fibrillation | through study completion, an average of 1 year
  Number of patients with a new onset of atrial fibrillation.
Vascular complications | through study completion, an average of 1 year
  Number of patients with major vascular complications.
Bleeding complications | through study completion, an average of 1 year
  Number of patients with life-threatening, disabling, or major bleeding complications.
Myocardial infarction | through study completion, an average of 1 year
  Number of patients with new myocardial infarction.
Acute kidney injury | up to 30 days post-procedure
  Number of patients with new onset of acute kidney injury stage II/III (AKIN classification).
Acute kidney injury | through study completion, an average of 1 year
  Number of patients with the need of renal replacement therapy.
New permanent pacemaker implantation | through study completion, an average of 1 year
  Number of patients with new permanent pacemaker implantation caused by new or worsened conduction disturbances.
Change in New York Heart Association (NYHA) classification | through study completion, an average of 1 year
  Severity of cardiac disease based on functional capacity will be described using the NYHA classification. Classification ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity.
Change in hemodynamic valve performance | through study completion, an average of 1 year
  Hemodynamic valve performance will be evaluated by echocardiography for aortic valve stenosis and aortic valve regurgitation (paravalvular & central).
Change in impairment caused by a stroke | through study completion, an average of 1 year
  Impairment caused by a stroke will be assessed using the the National Institutes of Health Stroke Scale (NIHSS)
Change in cognitive function | through study completion, an average of 1 year
  Cognitive function will be assessed using the Mini-mental state Examination-2 (MMSE-2) questionnaire
Change in the degree of disability in the daily activities | through study completion, an average of 1 year
  Degree of disability in the daily activities will be assessed using the modified Rankin Scale (mRS).
Change in Frailty Index | through study completion, an average of 1 year
  Frailty index will be assessed by the 5 Meter Walk Test, grip strength, Instrumental Activities of Daily Living and serum Albumin
Change in disease-specific health status | through study completion, an average of 1 year
  The health status in regards to congestive heart failure will be assessed by the patient using the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Change in health-related quality of life | through study completion, an average of 1 year
  The health-related Quality of Life will be assessed by the patient using The Medical Outcomes Study Short-Form 12 (SF-12) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Eltchaninoff, Prof., Principal Investigator — CHU Rouen - Hopital Charles Nicolle; Didier Tchétché, Dr., Principal Investigator — Clinique Pasteur Toulouse
Locations (48):
- Austria (4):
  - LKH-Univ. Klinikum Graz, Graz
  - Universitätskliniken Innsbruck, Innsbruck
  - Universitätsklinikum St. Pölten - Lilienfeld, Sankt Pölten
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (3):
  - Clinique Saint-Luc, Bouge
  - CHU De Charleroi, Charleroi
  - UZ Leuven Campus Gasthuisberg, Leuven
- Nicosia General Hospital, Nicosia, Cyprus
- Czechia (4):
  - University hospital Hradec Králové, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - IKEM (Institut Klinické a Experimentální Medicíny), Prague
  - Nemocnice Na Homolce, Prague
- Finland (2):
  - Helsinky University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (14):
  - CHU de Bordeaux - Hôpital cardiologique du Haut-Lévêqu, Bordeaux
  - CHRU de Brest, Brest
  - GHE-Hôpital Cardiologique Louis Pradel, Bron
  - CHU Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille - Institute Coeur Poumon, Lille
  - CHU Montpellier, Montpellier
  - CHU de Nantes - Hôpital Guillaume et René Laënnec, Nantes
  - Hôpital Privé Jacques Cartier, Paris
  - CHU et Université de Poitiers, Poitiers
  - CHU Rennes - Hopital de Pontchaillou, Rennes
  - CHU Rouen - Hopital Charles Nicolle, Rouen
  - Les Hopitaux Universitaires de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Frankfurt Am Main, Frankfurt
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- St. James´s Hospital, Dublin, Ireland
- Italy (6):
  - Azienda Ospedaliero Universitaria Policlinico "G.Rodolico - San Marco", Catania
  - A.O.U. Careggi, Florence
  - Ospedale del Cuore G. Pasquinucci, Massa
  - Universita di Padova, Padua
  - European Hospital, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (3):
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Leids Universitair Medisch Centrum, Leiden
  - St Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Switzerland (3):
  - Inselspital Universitätsspital Bern, Bern
  - Hirslanden Klinik Im Park, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Morriston Hospital, Morriston
  - Oxford University Hospitals - John Radcliffe hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva I, Alperi A, Hecht S, Zanuttini A, Theron A, Giuliani C, Camacho B, Dahou A, Mares J, Bax J, Bonaros N, Windecker S, Messika-Zeitoun D, Wesselink W, Rakova R, Bramlage P, Tchetche D, Eltchaninoff H, Pibarot P; RHEIA Trial Investigators. Echocardiographic Results of Transcatheter Versus Surgical Aortic Valve Replacement in Women With Severe Aortic Stenosis: The RHEIA Trial. J Am Heart Assoc. 2026 Jan 6;15(1):e047196. doi: 10.1161/JAHA.125.047196. Epub 2025 Dec 30. PMID 41467363
- [Derived] Tchetche D, Pibarot P, Bax JJ, Bonaros N, Windecker S, Dumonteil N, Nietlispach F, Messika-Zeitoun D, Pocock SJ, Berthoumieu P, Swaans MJ, Timmers L, Rudolph TK, Bleiziffer S, Leroux L, Modine T, van der Kley F, Auffret V, Tomasi J, Stastny L, Hengstenberg C, Andreas M, Leclercq F, Gandet T, Mascherbauer J, Trescher K, Prendergast B, Vasa-Nicotera M, Chieffo A, Mares J, Wesselink W, Rakova R, Kurucova J, Bramlage P, Eltchaninoff H. Transcatheter vs. surgical aortic valve replacement in women: the RHEIA trial. Eur Heart J. 2025 Jun 9;46(22):2079-2088. doi: 10.1093/eurheartj/ehaf133. PMID 40171878
- [Derived] Eltchaninoff H, Bonaros N, Prendergast B, Nietlispach F, Vasa-Nicotera M, Chieffo A, Pibarot P, Bramlage P, Sykorova L, Kurucova J, Bax JJ, Windecker S, Dumonteil N, Tchetche D. Rationale and design of a prospective, randomized, controlled, multicenter study to evaluate the safety and efficacy of transcatheter heart valve replacement in female patients with severe symptomatic aortic stenosis requiring aortic valve intervention (Randomized researcH in womEn all comers wIth Aortic stenosis [RHEIA] trial). Am Heart J. 2020 Oct;228:27-35. doi: 10.1016/j.ahj.2020.06.016. Epub 2020 Jun 30. PMID 32745733